CLINICAL TRIAL: NCT02096939
Title: Microvascular Function in Patients With Primary Aldosteronism and Essential Hypertension
Brief Title: Microvascular Function in Primary Aldosteronism
Status: Withdrawn | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Monica Schütten, MD, Maastricht University Medical Center
Other Study IDs: 48364
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Primary Aldosteronism; Essential Hypertension
MeSH Terms: conditions — Hyperaldosteronism; Essential Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Primary aldosteronism: Patients with primary aldosteronism, who undergo surgery or will be started on antihypertensive medication, including mineralocorticoid receptor antagonists
  Interventions: Procedure: Adrenal extirpation; Drug: Antihypertensive medication
- Essential hypertension: Patients with essential hypertension who will be started on antihypertensive medication
  Interventions: Drug: Antihypertensive medication

INTERVENTIONS:
Procedure: Adrenal extirpation
  Groups: Primary aldosteronism
Drug: Antihypertensive medication

SUMMARY:
Patients with primary aldosteronism, which is the most prevalent form of secondary hypertension, have an increased rate of cardiovascular events, compared to patients with essential hypertension, even with equal severity of hypertension. This might be partially attributed to the association of increased aldosterone levels with insulin resistance. How this relation can be explained from a pathophysiological point of view, is insufficiently established.

Recently, microvascular dysfunction has been proposed as a link between insulin resistance and hypertension. Loss of NO-mediated vasodilation is an important feature of microvascular dysfunction; in addition, an impaired insulin-mediated microvascular NO production has been suggested to underlie the reduction in insulin-stimulated glucose disposal that is characteristic of insulin-resistant states. Increased aldosterone levels are not only associated with insulin resistance, but also with endothelial dysfunction. In addition, they interfere with the vascular effects of insulin.

Therefore, the investigators hypothesize that in patients with primary aldosteronism, increased aldosterone levels induce microvascular dysfunction through reduction of NO-availability, which contributes to the development of insulin resistance, and of hypertension, in addition to the sodium-retaining effects of aldosterone.

ELIGIBILITY:
Inclusion Criteria:

Patients with primary aldosteronism

* Age 18-70 years
* Confirmed diagnosis of primary aldosteronism
* Serum potassium > 3.5 mmol/L with or without supplementation

Patients with essential hypertension

* Age 18-70 years
* Secondary causes of hypertension excluded

Exclusion Criteria:

* Cardiovascular disease (stroke, coronary artery disease, peripheral vascular disease, congestive heart failure, cardiac shunts, cardiac surgery, pulmonary hypertension, cardiac arrhythmias, family history of cardiac arrhythmias or sudden cardiac death)
* Diabetes mellitus
* Unstable or severe pulmonary disease
* Inflammatory diseases
* Alcohol use > 2 U/day (women) / > 3 U/day (men)
* (Frequent) use of acetylsalicylic acid, NSAID's, dipyridamole and corticosteroids
* eGFR < 60 mL/min
* Impairment of hepatic function
* Pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty patients with primary aldosteronism and twenty patients with essential hypertension
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Microvascular recruitment in skeletal muscle during hyperinsulinaemia | Baseline
Microvascular recruitment in skeletal muscle during hyperinsulinaemia | 3 months after (initiation of) treatment

CONTACTS AND LOCATIONS:
Overall Officials: Prof. C.D.A. Stehouwer, MD, PhD, Principal Investigator — Maastricht University Hospital